CLINICAL TRIAL: NCT04708990
Title: DELP for Acute Hemorrhagic Stroke: a Prospective, Random, Open-label, Blind-endpoint, Single Centre, Pilot Study
Brief Title: DELP for Acute Hemorrhagic Stroke
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: the research sponsors stopped further funding due to a planning of a multi-center trial
Sponsor: General Hospital of Shenyang Military Region (Other)
Responsible Party: Principal Investigator, Hui-Sheng Chen, Head of Neurology, General Hospital of Shenyang Military Region
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Y (2020) 044
Record Dates: First submitted 2021-01-11; First posted 2021-01-14 (Actual); Last update posted 2021-11-05 (Actual); Status verified 2021-10

CONDITIONS: Cerebral Hemorrhage
MeSH Terms: conditions — Cerebral Hemorrhage

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DELP (Experimental): Delipid Extracorporeal Lipoprotein filter from Plasma (DELP) is a non-pharmacological therapy for acute stroke, which is approved by China Food and Drug Administration
  Interventions: Device: Delipid Extracorporeal Lipoprotein filter from Plasma
- control group (No Intervention)

INTERVENTIONS:
Device: Delipid Extracorporeal Lipoprotein filter from Plasma — As a non-pharmacological therapy, Delipid Extracorporeal Lipoprotein filter from Plasma (DELP) hase been approved by China Food and Drug Administration to treat acute stroke
  Arms: DELP

SUMMARY:
Delipid Extracorporeal Lipoprotein filter from Plasma (DELP) has been found to improve neurological function and life ability of AIS patients and approved for the treatment of AIS by China Food and Drug Administration (CFDA). Our recent study imply that the neuroprotective effect of DELP involved multiple neuroprotective mechanism such as anti-inflammation, free radical scavenging, and decreasing MMP-9. Based on the multiple mechanisms, we argue that DELP may exert neuroprotective effect on acute cerebral hemorrhage.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-80;
* Spontaneous cerebral hemorrhage;
* Deep supratentorial intracerebral hemorrhage (basal ganglia and thalamus) with hematoma volume 5-40ml;
* NIHSS: 4-22;
* Time from onset to DELP is less than 48 hours;
* Premorbid mRS 0 or 1;
* Signed informed consent;

Exclusion Criteria:

* Secondary cerebral hemorrhage (secondary to trauma, tumor, vascular malformation, hemorrhage transformation of ischemic stroke, etc.);
* Comatose patients on admission (GCS score 3-8 on the Glasgow Coma Scale);
* Patients with intracerebral hemorrhage ruptured into the ventricle;
* Planed surgery;
* Severe hepatic or renal dysfunction, increase in ALT or AST (more than 2 times of upper limit of normal value), increase in serum creatinine (more than 1.5 times of upper limit of normal value) or requiring dialysis;
* Severe hypertension (systolic blood pressure over 200mmHg or diastolic blood pressure over 110 mmHg);
* Previous allergy to heparin or calcium;
* hypoproteinemia;
* Unsuitable for this clinical studies assessed by researcher.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-01-12 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with modified Rankin Score 0 to 2 | Day 90

SECONDARY OUTCOMES:
Proportion of patients with modified Rankin Score 0 to 1 | Day 90
Changes in national institutes of health stroke scale (NIHSS) | 48 hours
  NIHSS ranges from 0-42, and the decrease in NIHSS means the improvement of neurological deficit.
changes of hematoma volume compared with the baseline | 48 hours
changes of edema volume around hematoma compared with the baseline | 48 hours
the occurence of death due to any cause | Day 90

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurology, General Hospital of Northern Theater Command, Shenyang, China